CLINICAL TRIAL: NCT05324995
Title: Comparing Pre-emptive Injection of Peri-Articular-Multimodal Drug With Oral Celecoxib for Postoperative Pain Management in Total Knee Arthroplasty: A Randomized Clinical Trial
Brief Title: Peri-Articular-Multimodal Drug and Oral Celecoxib in Management of Postoperative Pain of Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Shafa, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 394048
Record Dates: First submitted 2022-01-08; First posted 2022-04-13 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain; Total Knee Arthroplasty
Keywords: Total knee arthroplasty; Pain; Multimodal analgesia; Range of motion
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Epinephrine; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigator who performed the baseline and follow-up assessments and the patients were unaware of the study group; as the investigator was absent at the time of the surgery and all the patients administered a pill prior to the surgical procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multimodal injection (Experimental): The first group was treated using a preemptive periarticular injection of multimodal drugs. Therefore, a combination of drugs consisted of 50 mg bupivacaine hydrochloride 0.5% (AstraZeneca, Cenexi, France), 1 ml morphine sulfate 10 mg/ml (DarouPakhsh, Tehran, Iran), 300 mcg epinephrine (1:1000) (DarouPakhsh, Tehran, Iran) and 30 mg ketorolac (Caspian Tamin, Rasht, Iran) diluted by 0.9% sodium chloride solution to make a total 100 ml of injection drug was injected in periarticular area. The injections were done within 15 minutes before the incision in seven areas of the joint as followed: 15 ml in posterolateral soft tissue and lateral femoral periosteum, 15 ml posteromedial soft tissue and medial femoral periosteum, 20 ml inferomedial capsule, 20 ml superomedial capsule, 10 ml lateral capsule, 10 ml medial subcutaneous tissues and 10 ml lateral subcutaneous tissue.
  Interventions: Drug: Multimodal Drug
- epinephrine group (placebo group) (Experimental): The second group received 300 mcg epinephrine (1:1000) (DarouPakhsh, Tehran, Iran) peri-articulary, similar to the first group.
  Interventions: Drug: epinephrine
- celecoxib group (control group) (Experimental): The third group administered celecoxib (200 mg) orally immediately before the surgery initiation.
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: Multimodal Drug — The Multimodal Drug group received morphine, epinephrine, and ketorolac (n=48), The epinephrine group (placebo group) (n=49) received 300 mcg epinephrine (1:1000) (DarouPakhsh, Tehran, Iran) peri-articulary,and the celecoxib group(control group)(n=49) recieved 400mg celecoxib orally
  Other Names: Case
  Arms: Multimodal injection
Drug: epinephrine — The second group received 300 mcg epinephrine (1:1000) (DarouPakhsh, Tehran, Iran) peri-articulary
  Other Names: Placebo
  Arms: epinephrine group (placebo group)
Drug: celecoxib — The third group administered celecoxib (200 mg) orally immediately before the surgery
  Other Names: Control
  Arms: celecoxib group (control group)

SUMMARY:
This study is a randomized-clinical-trial on 146 patients candidate for total knee arthroplasty (TKA) who were randomly allocated to three treatment groups, including 1) a cocktail consisting of bupivacaine, morphine, epinephrine, and ketorolac (n=48), 2) only epinephrine (placebo group) (n=49), and 3) 400mg celecoxib orally (control group) (n=49) using Random Allocation software. The injections and oral therapy were performed within 15 minutes before the surgical procedure. The study's primary outcome was the Knee Society Score (KSS) calculated at baseline, within six weeks and six months postoperatively. Range of motion (ROM) and Visual Analogue Scale (VAS) to assess pain intensity as the other primary outcomes were evaluated before the procedure, within 24 hours, 48 hours, and six weeks postoperatively.

DETAILED DESCRIPTION:
This randomized clinical trial conducted on 146 patients undergone TKA in orthopedic hospitals affiliated at Isfahan University of Medical Science (IUMS) in 2021.

The presence of osteoarthritis, making the patients candidate for primary unilateral total knee arthroplasty (TKA), and body mass index of 20-30 kg/m2 were determined as inclusion criteria.

The Regional Bioethics Committee of IUMS approved the study protocol. This study was designed as a census study; therefore, all the patients who met the criteria for participation in this study were recruited. Participants were randomly divided into three groups using Random Allocation software, so each patient was provided with a specific number from 1-to-146 by the software and allocated to one of the groups.

The investigator who performed the baseline and follow-up assessments and the patients were unaware of the study group; as the investigator was absent at the time of the surgery and all the patients administered a pill prior to the surgical procedure (one group was treated with celecoxib and the other two ones administered placebo similar in shape and color with celecoxib).

The primary outcome was the Knee Society Score (KSS) calculated at baseline, within six weeks and six months postoperatively. Range of motion (ROM) and Visual Analogue Scale (VAS) to assess pain intensity as the other primary outcomes were evaluated before the procedure, within 24 hours, 48 hours, and six weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoarthritis
* Candidate for primary unilateral TKA
* Body mass index of 20-30 kg/m2

Exclusion Criteria:

* Unable to follow-up the assessments
* Having more than 20% defects in medical records

Ages: 37 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Baseline Measurements of Knee Society Score (KSS) | At the beginning of the study
  The Knee Society score is an assessment of the knee that comprises two arms, the functional ability and clinical examination scores, each with a 100-point denominator. One-hundred points are allocated to the functional capacity, including walking distance, stair-climbing ability, and the use of walking aids.
Baseline range of motion (ROM) | At the beginning of the study
  Knee ROM was evaluated using a standard goniometer
visual analogue scale (VAS) | 24 hours after the surgical procedure
  Visual Analogue Scale (VAS) was used to evaluate the patient's postoperative pain intensity with a 0 to 10 rating scoring scale
Range of motion (ROM) | 6 months after surgery
  Knee ROM was evaluated using a standard goniometer
Knee Society Score (KSS) | 6 months after surgery
  The Knee Society score is an assessment of the knee that comprises two arms, the functional ability and clinical examination scores, each with a 100-point denominator. One-hundred points are allocated to the functional capacity, including walking distance, stair-climbing ability, and the use of walking aids.
visual analogue scale (VAS) | 48 hours after the surgical procedure
  Visual Analogue Scale (VAS) was used to evaluate the patient's postoperative pain intensity with a 0 to 10 rating scoring scale
visual analogue scale (VAS) | Six weeks after surgery
  Visual Analogue Scale (VAS) was used to evaluate the patient's postoperative pain intensity with a 0 to 10 rating scoring scale

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
It is confirmed to IPD be shared with other researchers
Supporting Information: Study Protocol, CSR
Time Frame: After getting the code
Access Criteria: No limitation